CLINICAL TRIAL: NCT00821730
Title: Exploring the Learning Needs of Individuals With Inflammatory Arthritis From the Perspectives of Patients, Family Members and Friends, and Health Care Providers: Perspectives of Family Members and Friends
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University of Toronto (Other); University Health Network, Toronto (Other)
Responsible Party: Dr. Mary J. Bell, Division of Rheumatology, Sunnybrook Health Sciences Centre
Other Study IDs: DOCH2 446-2008
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Early Inflammatory Arthritis
Keywords: Mixed methods research (qualitative and quantitative); Peer support; Early inflammatory arthritis; Self-management; Patient education
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Biospecimen Retention: None Retained — This is a qualitative research study
Oversight: Data Monitoring Committee: No

SUMMARY:
nflammatory arthritis (IA) is a major cause of long-term disability. Due to specialist shortages, failure of primary care providers and individuals to recognize the disease, and lack of awareness of the importance of early intervention, delays to rheumatologic care are common. Peer support models have been used for various health issues and may be one method to assist individuals with early IA to manage their disease and cope with stress. One-on-one semi-structured interviews will seek out feedback on a peer support approach and explore the learning needs (informational needs, educational preferences) and opinions about emotional and appraisal support of individuals living with IA from the perspectives of family and friends. The data will be analyzed and expressed themes (articulated needs and understandings of interviewee context) will guide the future development of a peer support intervention.

DETAILED DESCRIPTION:
I. Rationale

Inflammatory arthritis is one of the most prevalent diseases in Canada, affecting about 10% of Canadian adults (Health Canada, 2003). It is a leading cause functional disability, chronic pain, and reduced quality of life, resulting in difficulties at work and at home. Affected individuals experience general malaise and fatigue, persistent morning stiffness, and severe joint pain. Also, the course and symptoms of the disease over time are often unpredictable, making management difficult (Smolen and Aletaha, 2005).

Currently, there is no clear etiology for inflammatory arthritis, nor is there a definitive cure. Existing treatments have been shown to maintain daily function, delay onset of disability and alleviate pain. These include traditional medical treatment such as nonsteroidal anti-inflammatory drugs (NSAIDs), low-dose oral glucocorticoids, disease modifying anti-rheumatic drugs (DMARDs), and biologic agents to control local inflammatory processes (Altman et al., 2000; American College of Rheumatology, 2002). Although medications for self-care of patients are important, both educational programs and peer support have played historic yet vital roles in helping individuals with inflammatory arthritis better cope with their disease (Penninx et al., 1997; Tucker and Kirwan, 1991)

Early treatment is of particular importance for patients diagnosed with inflammatory arthritis. One way to ensure prompt treatment to these patients is to enhance knowledge and skills of both patients and their caregivers in order to improve decision-making and help individuals manage disease. Patient education can help individuals and their family members with patient self-care and prepare them to make decisions regarding their treatment (Koehn and Esdaile, 2008). Also, better understanding of the relationship between clinical practice and patient- and family-perceived needs will result in better patient-centered care (Koehn and Esdaile, 2008).

It is widely recognized that peer support plays a key role in the treatment of any disease (Berkman et al., 2000). These social support groups include the family members and friends of individuals with disease who can help them with treatment decisions and provide emotional support while they cope with their disease. In general, having social support leads to positive impact on quality of life (Savelkoul and de Witte, 2001) whereas lacking high quality social relationships may lead to anxiety, depression, loneliness, and poor physical health (Berkman et al., 2000).

There is extensive literature exploring both peer support and patient education and their associations with arthritis. Recent studies have revealed that individuals newly diagnosed with rheumatoid arthritis look for not only informational support about symptoms and management, but also emotional support such as having someone or a group to talk to (Radford et al., 2008). Sherman (2003) reported that peer support provides happiness and boosts self-esteem in patients with knee osteoarthritis. Patient education has been shown to increase compliance with leisurely physical activity in individuals with rheumatoid arthritis (Mayoux-Benhamou et al., 2008). Group sessions including partners of patients with inflammatory arthritis have led to mixed results regarding the effectiveness of spousal participation (Martire et al., 2008; van Lankveld W, 2004; Riemsma et al., 2003). Less is known about the specific educational needs of family members and friends of individuals newly diagnosed with inflammatory arthritis.

II. Purpose and Objectives

The purpose of this study is to explore the learning needs of individuals with inflammatory arthritis from the perspective of family members and friends of those with inflammatory arthritis. In particular, this study aims to explore the types of support patients and their families feel would be most helpful upon diagnosis. Specific objectives of this study include:

* to examine the learning preferences of family members and friends of individuals who have inflammatory arthritis, including thoughts about peer support,
* to identify specific informational needs related to managing arthritis, and
* to explore how learning needs change over time or duration of the disease.

Objectives will be addressed through semi-structured interviews of family members and friends of patients through the Sunnybrook Health Sciences Centre rheumatology clinic.

III. Methodology

In order to meet these objectives, the perspectives of family members and friends of individuals with inflammatory arthritis will be explored using a qualitative approach. In particular, semi-structured interviews will be used.

III. A. Semi-structured Interviews

Study Design Semi-structured interviews will be conducted with key informants, defined as individuals who have good knowledge and understanding about the disease of their family member or friend with inflammatory arthritis and can clearly articulate their knowledge. These interviews serve as an investigative technique for gathering data in short period of time and to gain new insight and a broad perspective of views on the research question. Although the same specific questions will be asked in the same manner with each interview, the interviewer will be free to alter the order in which questions are asked so that the interview caters towards each individual research participant. An interview guide (Appendix A) was developed for the purpose of this study, and an interview notes form (Appendix B) will be used for interviews. As it is a semi-structured interview approach, certain probe questions that aim to encourage research participants to elaborate on their responses and further discussion have not been included in this guide. Such probe questions are context-dependent and evolve as the interview takes place.

Detailed field notes will be recorded during and after each interview, using the interview notes form (Appendix B) as a guide. Digital recorders will be used to record interviews. All digital audio files will be transcribed verbatim. All field notes and digital audio files will be uploaded to NVivo8, a qualitative data management software serving to assist in the analysis, synthesis, and management of data. Data transcription will be outsourced. A data transfer agreement will be put in place with Sunnybrook Research Administration.

Data will be interpreted after each interview. Additional questions may be added to the interview guide for subsequent interviews. Data will be collected until approximately 10 to 15 research participants are interviewed, or until there is enough information gathered such that saturation of data is obtained - i.e., no new concepts arise from the data.

Each interview is anticipated to last approximately one hour, and will conducted by a second-year medical student trained by the study coordinator who has expertise in qualitative research.

Subjects

Potential research participants will be identified for participation in this study based on the following inclusion criteria:

* Participants must be a family member or a care-giving friend of an individual diagnosed with inflammatory arthritis by an established physician;
* Participants must be aged 18 years or older;
* Participants must be able to participate in a 1 hour interview; and
* Participants must be able to understand and converse in English.

Recruitment and Consent Process

Individuals will be identified by Dr. Mary Bell (Principal Investigator) through her rheumatology clinic at Sunnybrook Health Sciences Centre. A flyer (Appendix H) will be given to the patient by the PI to pass on to their friends or family members which would include information about the study and how to contact the study team if they are interested in participating. Upon contacting the study team, Dr. Bell will identify and screen family members of patients according to the eligibility criteria for the study and will initiate the informed consent process (Appendix C). Dr. Bell will then introduce the project and review both an information letter (Appendix D) on the study and a consent form (Appendix C) with each eligible patient. This will be done to ensure that each potential research participant understands the purpose of the study and what is being asked of them. When an individual has verbally agreed to participate, his/her name will be forwarded to the Office Manager at the clinic who will contact the individual and schedule an interview at Dr. Bell's rheumatology clinic office with the medical student co-investigator assigned to the project. A confirmation letter (Appendix E) on a Sunnybrook Health Sciences Centre letterhead signed by Dr. Bell will be mailed to the potential research participant; this will include the time and location of the interview. One day prior to the scheduled interview, the medical student will telephone the individual to remind them of the time and location of the interview using a standardized telephone script (Appendix F). At the beginning of the interview, prior to asking any questions, the medical student will review the consent form, answer any further questions the person may have and subsequently obtain written consent from the individual prior to commencing the interview. Once written consent is obtained, a copy will be provided to the research participant.

IV. Data Analysis

A constant comparative method (Strauss and Corbin, 1998) will be used to describe learning needs using open-coding methods. Transcripts from each interview will independently categorized by two members of the research team. Each team member will first analyze the data independently before meeting to compare and come to an understanding of common emergent themes that may arise during interviews. Each transcript will be compared and consensus reached as to the code to assign a particular unit of text. A coding scheme will evolve as data analysis progresses and themes will be derived through synthesis.

V. Risks and Benefits

There are no known risks associated with this study. Participants of interviews may benefit from having any questions they may have answered off-the-record before or after interviews. Potential indirect benefits include improvement in care provided to individuals with inflammatory arthritis, particularly from the perspective of their family members and friends, and the opportunity to share their experiences with other family members or friends of individuals with inflammatory arthritis.

VI. Privacy and Confidentiality

Only the Principal Investigator and the members of the research team who conduct interviews will know the identity of research participants. Confidentiality will be ensured by assigning each research participant a unique identifying number upon agreeing to participate in the study. The list of names, addresses, and phone numbers corresponding to each study number and all other identifying information will be kept on password-protected computers on a secure server in a locked research room. All information obtained during the study will be held in strict confidence, and any electronic data will be password-protected and stored on a secure server in a locked research room. No names or identifying information will be used in any publications or presentations, nor will they be transferred outside researchers in this study. All hard copies of data will be stored in a locked research room at the Sunnybrook Health Sciences Centre. Data will be retained for 25 years as stated in the protocol and informed consent form.

VI. Compensation

No monetary remuneration will be provided. However, transportation costs will be covered (e.g., subway tokens, taxi fares, parking) and refreshments will be provided (see Appendix G for budget).

VIII. Communication of Results

Results from this study will be disseminated to research participants. Results will be communicated to an academic and health professional audience through scientific publications and presentations of findings. No identifying information will be contained in these reports or presentations. All results presented will be in keeping with privacy and confidentiality issues as addressed in section VI.

A presentation based on findings will be given to second year medical students at the University of Toronto. Information given within the presentation will be shared with the course coordinators of the Determinants of Community Health Year 2 course under the Faculty of Medicine at the University of Toronto. Reports will be made available upon request.

ELIGIBILITY:
Inclusion criteria

* Participants must be a family member or a care-giving friend of an individual diagnosed with inflammatory arthritis by an established physician;
* Participants must be aged 18 years or older;
* Participants must be able to participate in a 1 hour interview; and
* Participants must be able to understand and converse in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family members, caregivers and friends of individuals with inflammatory arthritis
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Bell, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada